CLINICAL TRIAL: NCT02820337
Title: ObéVIH : Pathophysiology of Adipose Tissue of Obese HIV-infected Patients Undergoing a Sleeve Gastrectomy Using Single Port
Brief Title: Pathophysiological Study of Adipose Tissue of Patients Infected With HIV
Acronym: ObéVIH
Status: Completed | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 05
Record Dates: First submitted 2016-04-29; First posted 2016-06-30 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- non comparative: Bariatric surgery patients infected with HIV, overweight with controlled viral load and HIV lipohypertrophy particularly truncal

SUMMARY:
The main goal of our project is the study of subcutaneous and visceral (SAT and VAT) adipose tissue taken during bariatric surgery (Single port sleeve gastrectomy) of subjects with HIV infection, anf morbid obesity with undetectable viral load (VL) and having HIV lipohypertrophy particularly truncal. The study covers both the morphology of adipocytes,fibrosis, immune activation and inflammation, gene expression, pharmacology of antiretroviral drugs (ARV) and the measurement of viral replication in the adipose tissue and the plasma before and after bariatric surgery.

DETAILED DESCRIPTION:
The choice of the sleeve gastrectomy is based on choosing an effective technique with few complications, no rupture of digestive continuity and therefore little malabsorptive effect with a better quality of life.

The intervention of sleeve gastrectomy offers a unique opportunity to study the SAT and VAT of HIV obese patients before and after bariatric surgery, to analyze the specific modifications of this tissue and to better understand the pathophysiology of this disease. The term associated with changes in cardiometabolic comorbidities and their improvement after weight loss will be important elements in the management of these patients. It is therefore important to evaluate whether the fibrosis term changes observed in HIV patients will change the effectiveness of the intervention.

In the general population, obesity is a major public health problem. It is considered an inflammatory disease, multifactorial with chronic evolution, which requires long-term medical care and / or surgery . Indeed, the body mass index (BMI) correlates with increased mortality mainly due to cardiovascular diseases (hypertension, coronary artery disease), cancer and diabetes. Finally, overweight and obesity are the leading causes of liver disease in Western countries resulting in nonalcoholic fatty liver disease, a term that includes all the hepatic lesions observed in overweight and obesity: steatosis, steatohepatitis, fibrosis, cirrhosis or hepatocellular carcinoma. Nonalcoholic fatty liver disease reflects not only the presence of insulin resistance but also participates in its installation. Reducing overweight is therefore a key part of treatment to reduce chronic inflammation, insulin resistance and liver damage.

There is little data in the literature on the prevalence of obesity in the population of HIV patients. In France, the prevalence of obesity in the French Hospital Database on HIV is 15.1% among women and 5.3% among men, similar to prevalence in the general population. Patients born in sub-Saharan Africa have a higher risk with 20.7% versus 12.2% in women and 10.9% versus 4.7% for men.

No data is available on the obesity complications described in the general population in our population of obese HIV patients. Nevertheless, apart from obesity, patients infected with HIV develop cardiovascular and metabolic complications well documented in recent years.

French and international recommendations agree that the management of obesity should be multidisciplinary. In the treatment, surgical treatment is the treatment of choice in French and international recommendations in the following indications:

* morbid obesity (BMI ≥ 40 kg / M²) resistant to medical treatment and exposing patients to serious complications that can not be controlled by the specific treatment
* obesity with BMI between 35 and 40 kg / M² with comorbidities associated with life-threatening or functional outcomes: cardiovascular disease, musculoskeletal disease, severe metabolic disorders not controlled by maximal medical therapy. In each case, the indication can be considered in patients who have had access to specialized medical care for at least 6 months, also including complementary approaches (diet, physical activity, management of psychological problems, treatment complications).

At present, the sleeve gastrectomy is the technique of choice in the general population with, compared to other bariatric surgery techniques such as bypass, reducing complications, length of hospital stay, operative time, a gain in term quality of life without disruption of digestive continuity and therefore little or no malabsorption. This lack of malabsorption it an argument of choice in our HIV patients on cART with a reduced risk of malabsorption of ARV and vitamin deficiencies such as vitamin D deficiency already well described in HIV. The minimally invasive approach (1 trocar), routinely performed by Dr. G. Pourcher for obese patients whether they are infected with HIV, reduces surgical risk. This Single port also allows easy access to SAT, VAT and liver.

The management of obesity in the HIV population, now having a similar life expectancy should be the same as that of the general population but remains to this day very marginal. The literature on the subject is almost "poor" Additionally, comorbid conditions existing in the population of HIV patients are a target population requiring support at least equivalent to that of the general population.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection,
* Aged to 18 at 65 ans,
* Obesity defined as a Body Mass Index (BMI)> 35 kg / M² with comorbidities Or BMI > 40 kg/M²
* Forget bariatric surgery after a positive opinion of the specialized multidisciplinary meeting
* on stable antiretroviral therapy for 12 months
* with controlled HIV infection (<50 copies / ml)
* Signed informed consent
* Karnofsky Index > 80 %
* Patient affiliated or beneficiary of a national insurance scheme (article L1121-11 of the Public health code) (the Medical aid of State or SOUL is not a national insurance scheme)

Exclusion Criteria:

* Uncontrolled severe infection
* Current pregnancy (positive HCG)
* Saving justice, guardianship
* Participation to another study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathophysiology of adipose tissue of obese HIV-infected patients undergoing a sleeve gastrectomy using single port.
  20 patients will be required. Patients will be included after positive opinion of the multidisciplinary meeting of management of obesity.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Measure of fibrotest to assess the liver fibrosis | 30 months
  fibrotest is the estimated index of liver fibrosis established according to the assay values of 5 parameters: alpha-2 macroglobulin, haptoglobin, apolipoprotein-A1, total bilirubin and g-glutamyl-transpeptidase.
Measure of actitest to assess the liver inflammation | 30 months
  ActiTest gives an estimate of the intensity of the inflammation and liver cell killing activity. ActiTest uses 5 markers fibrotest which is added the dosage of transaminases measure of Ambulatory blood pressure.
Measure of steatotest to assess the liver steatosis | 30 months
Measure of serum inflammatory biomarkers assessed by ELISA assay | 30 months
Measure of viral load in plasma and adipose tissue assessed by quantification using Cobas 6800 system/cobas HIV-1 Test (Roche) | 30 months
Measure of the pharmacokinetics of antiretrovirals by estimating trough plasma concentrations using mass spectrometry assay. | 30 months
Measure of the pharmacokinetics of antiretrovirals by estimating trough adipose tissue concentrations using mass spectrometry assay. | 30 months

SECONDARY OUTCOMES:
Measure of left ventricular mass assessed by echocardiography to evaluate cardiovascular function | 30 months
Measure of Volume of epicardial fat assessed by echocardiography to evaluate cardiovascular function | 30 months
Carotid intima media thickness assessed by echo-doppler to evaluate cardiovascular atherosclerosis | 30 months
Score of calcification assessed by cardiac CT to evaluate cardiovascular atherosclerosis | 30 months
Measure of body composition assessed by dexascan to evaluate the impact of sleeve gastrectomy | 30 months
Measure of the surface of the adipose tissue subcutaneous and visceral assessed by tomodensitometry to evaluate the impact of sleeve gastrectomy | 30 months
Measure of bone mineral density assessed by dexascan to evaluate the impact of sleeve gastrectomy | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Valérie POURCHER MARTINEZ, MD, PhD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Yasmine Dudoit, Paris, France

IPD SHARING:
Plan to Share IPD: No